CLINICAL TRIAL: NCT01916070
Title: Syncope Patient Evaluation in the Emergency Department (SPEED)
Brief Title: Syncope Patient Evaluation in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Christ, Prof. Dr. med. Michael Christ, Klinikum Nürnberg
Other Study IDs: SPEED01
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: (Near) Syncope
Keywords: syncope; near syncope; prognosis; emergency department
MeSH Terms: conditions — Syncope; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with syncope
- patients with near syncope

SUMMARY:
Patients with the symptom complex syncope or near-syncope are quite often in the emergency department. Most patients with syncope have a positive prognosis. However some types of syncope are associated with an increased morbidity and mortality. It is a challenge to detect these patients reliably at an early stage. The current guidelines contain exact definitions concerning the characteristics of patients with syncope and recommendations on how to diagnose and treat these patients following standardized pathways. Due to the fact that near-syncope is poorly defined and therefore seldom evaluated in clinical trials, data concerning near-syncope are rare.

Our aim was to characterize patients presenting with syncope or near-syncope to the emergency department regarding their risk profile, comorbidities and prognosis. First we evaluated if there is a difference between the two groups syncope and near-syncope concerning type and frequency of adverse events. Furthermore we analyzed the routinely measured cardiac biomarkers NT-proBNP and hs cTnT in patients with syncope or near-syncope. Then we determined both their prognostic accuracy in predicting adverse events and their diagnostic accuracy in finding the underlying etiology. Finally we analyzed a special patient collective, patients aged ≥ 65 years. It is assumed that elderly patients are suffering from comorbidities and age-related physiological and cognitive disabilities. We therefore hypothesize that elderly patients, in contrast to patients aged < 60, display an increased risk of adverse events and that they have a poorer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* (near) syncope

Exclusion Criteria:

* age < 18 years
* progressive impairment of consciousness
* use of mind-altering drugs
* non syncopal loss of consciousness: hyperventilation, hypoglycaemia, metabolic disorders, psychogenic pseudosyncope, TIA or stroke, seizure, transient loss of consciousness caused by craniocerebral injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with (near) syncope to the emergency department
Sampling Method: Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
adverse events in patients with syncope and near syncope within 30 days after presentation to the emergency department | 30 days

SECONDARY OUTCOMES:
prevalence and prognosis of patients with syncope or near syncope in the emergency department | 6 months
prognostic and diagnostic accuracy of cardiac biomarkers NTproBNP and hs-cTnT | 6 months
prevalence, prognosis and clinical assessment of elderly patients ≥ 65 years with (near) syncope in the emergency department | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Christ, Prof., Principal Investigator — Klinikum Nürnberg
Locations (1):
- Klinikum Nuremberg, Nuremberg, Bavaria, Germany